CLINICAL TRIAL: NCT04682756
Title: A Multicenter Study on Early Diagnosis of NSTE-ACS Patients Based on Machine Learning Model
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Xinjiang Medical University (Other)
Collaborators: Shihezi University (Other)
Responsible Party: Principal Investigator, Xiang Ma, Department of Cardiology, First Affiliated Hospital of Xinjiang Medical University
Other Study IDs: XMa
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: NSTEMI - Non-ST Segment Elevation MI; Unstable Angina
Keywords: NSTEMI; UA; Machine Learning
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CNN model: Electronic health information of NSTEMI and UA patients in two chest pain centers from 2017 to 2019 was collected，After manual labeling, the characteristics of patient admission records were selected, and through the construction of one-dimensional convolution (CNN) model. Taking the multi-fold cross-validation and ROC-AUC curve as the measurement index, 75% of the data are modeled and 25% of the data are used to verify the effect of the model.
  Interventions: Diagnostic Test: The model of machine learning
- XG boost: Through the construction of XG boost model,taking the multi-fold cross-validation and ROC-AUC curve as the measurement index, 75% of the data are modeled and 25% of the data are used to verify the effect of the model.
  Interventions: Diagnostic Test: The model of machine learning

INTERVENTIONS:
Diagnostic Test: The model of machine learning — Early diagnosis of NTEMI patients by machine learning model

SUMMARY:
Early diagnosis of NSTEMI and UA patients is mainly through the construction of machine learning model.

DETAILED DESCRIPTION:
The patients with NSTEMI and UA were included. After manual labeling, the admiss- ion record characteristics of patients were selected. 75% of the data is used to build the model, and 25% of the data is used to verify the validity of the model. Five classification models of one-dimensional convolution (CNN), naive Bayesian (NB), support vector machine (SVM), random forest (RF) and ensemble learning were constructed to identify and diagnose NSTEMI and UA patients. Multi-fold cross-validation and ROC-AUC curve are used to measure the advantages and disadvantages of the models.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included and excluded strictly according to the diagnostic criteria of Chinese guidelines for diagnosis and treatment of Non-STsegment elevation acute coronary syndrome (2016). The patients were admitted to the hospital with chest pain as the main complaint, and were admitted to the first affiliated Hospital of Xinjiang Medical University and the first affiliated Hospital of Medical College of Shihezi Univ- ersity. the patients were diagnosed as NSTEMI and UA by coronary angiography (age range from 30 to 75 years old).

Exclusion Criteria:

- 1. Patients with STEMI, aortic dissecting aneurysm, pneumothorax and other non-cardiogenic chest pain. 2.Severe hepatorenal failure, primary tumor without surgical treatment, non-severe infection complicated with shock and pregnant women. 3.Previous severe valvular disease, viral myocarditis, pericardial effusion, cardiac pacemaker implantation, cardiogenic shock with serious complications, hypertensive heart disease, various cardiomyopathy, congenital heart disease, etc.

4.Patients with heart disease, AECOPD, lung tumor and hyperthyroidism were diagnosed in the past.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with NSTEMI and UA were included in the Chest Pain Center of the First Affiliated Hospital of Xinjiang Medical University and the First Affiliated Hospital of Medical College of Shihezi University from 2017 to 2019.
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Accurate diagnosis of NSTEMI from patients with acute chest pain | Within 1 year
  NSTEMI patients are accurately diagnosed from patients with acute chest pain through a trained machine learning algorithm. Our model uses multi-fold cross-validation and ROC-AUC curve as the measurement index, 75% of the data are modeled, and 25% of the data verify the effect of the model. For this reason, we will calculate the accuracy, specificity and likelihood ratio when the sensitivity cutoff value is 0.9.

CONTACTS AND LOCATIONS:
Overall Officials: Aikeliyaer Ainiwaer, M.D, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Quan Qi, Ph.D, Study Director — College of Information and Technology, Shihezi University; Yi Ying Du, M.D, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University
Locations (1):
- The first affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Machine learning model to identify patients with UA and NSTMI

REFERENCES:
- [Background] Cuocolo R, Perillo T, De Rosa E, Ugga L, Petretta M. Current applications of big data and machine learning in cardiology. J Geriatr Cardiol. 2019 Aug;16(8):601-607. doi: 10.11909/j.issn.1671-5411.2019.08.002. PMID 31555327
- [Background] Ambale-Venkatesh B, Yang X, Wu CO, Liu K, Hundley WG, McClelland R, Gomes AS, Folsom AR, Shea S, Guallar E, Bluemke DA, Lima JAC. Cardiovascular Event Prediction by Machine Learning: The Multi-Ethnic Study of Atherosclerosis. Circ Res. 2017 Oct 13;121(9):1092-1101. doi: 10.1161/CIRCRESAHA.117.311312. Epub 2017 Aug 9. PMID 28794054
- [Background] Weng SF, Reps J, Kai J, Garibaldi JM, Qureshi N. Can machine-learning improve cardiovascular risk prediction using routine clinical data? PLoS One. 2017 Apr 4;12(4):e0174944. doi: 10.1371/journal.pone.0174944. eCollection 2017. PMID 28376093
- [Background] Patel BB, Sperotto F, Molina M, Kimura S, Delgado MI, Santillana M, Kheir JN. Avoidable Serum Potassium Testing in the Cardiac ICU: Development and Testing of a Machine-Learning Model. Pediatr Crit Care Med. 2021 Apr 1;22(4):392-400. doi: 10.1097/PCC.0000000000002626. PMID 33332868
- [Background] Groepenhoff F, Eikendal ALM, Bots SH, van Ommen AM, Overmars LM, Kapteijn D, Pasterkamp G, Reiber JHC, Hautemann D, Menken R, Wittekoek ME, Hofstra L, Onland-Moret NC, Haitjema S, Hoefer I, Leiner T, den Ruijter HM. Cardiovascular imaging of women and men visiting the outpatient clinic with chest pain or discomfort: design and rationale of the ARGUS Study. BMJ Open. 2020 Dec 15;10(12):e040712. doi: 10.1136/bmjopen-2020-040712. PMID 33323438
- [Background] Kwon JM, Jeon KH, Kim HM, Kim MJ, Lim S, Kim KH, Song PS, Park J, Choi RK, Oh BH. Deep-learning-based risk stratification for mortality of patients with acute myocardial infarction. PLoS One. 2019 Oct 31;14(10):e0224502. doi: 10.1371/journal.pone.0224502. eCollection 2019. PMID 31671144
- [Background] Chowdhury MEH, Alzoubi K, Khandakar A, Khallifa R, Abouhasera R, Koubaa S, Ahmed R, Hasan MA. Wearable Real-Time Heart Attack Detection and Warning System to Reduce Road Accidents. Sensors (Basel). 2019 Jun 20;19(12):2780. doi: 10.3390/s19122780. PMID 31226858
- [Background] Wu CC, Hsu WD, Islam MM, Poly TN, Yang HC, Nguyen PA, Wang YC, Li YJ. An artificial intelligence approach to early predict non-ST-elevation myocardial infarction patients with chest pain. Comput Methods Programs Biomed. 2019 May;173:109-117. doi: 10.1016/j.cmpb.2019.01.013. Epub 2019 Jan 31. PMID 31046985
- [Background] Bernatz S, Ackermann J, Mandel P, Kaltenbach B, Zhdanovich Y, Harter PN, Doring C, Hammerstingl R, Bodelle B, Smith K, Bucher A, Albrecht M, Rosbach N, Basten L, Yel I, Wenzel M, Bankov K, Koch I, Chun FK, Kollermann J, Wild PJ, Vogl TJ. Comparison of machine learning algorithms to predict clinically significant prostate cancer of the peripheral zone with multiparametric MRI using clinical assessment categories and radiomic features. Eur Radiol. 2020 Dec;30(12):6757-6769. doi: 10.1007/s00330-020-07064-5. Epub 2020 Jul 16. PMID 32676784
- [Background] Md Idris N, Chiam YK, Varathan KD, Wan Ahmad WA, Chee KH, Liew YM. Feature selection and risk prediction for patients with coronary artery disease using data mining. Med Biol Eng Comput. 2020 Dec;58(12):3123-3140. doi: 10.1007/s11517-020-02268-9. Epub 2020 Nov 6. PMID 33155096
- [Background] Allen B, Molokie R, Royston TJ. Early Detection of Acute Chest Syndrome Through Electronic Recording and Analysis of Auscultatory Percussion. IEEE J Transl Eng Health Med. 2020 Sep 30;8:4900108. doi: 10.1109/JTEHM.2020.3027802. eCollection 2020. PMID 33094035
- [Background] Eberhard M, Nadarevic T, Cousin A, von Spiczak J, Hinzpeter R, Euler A, Morsbach F, Manka R, Keller DI, Alkadhi H. Machine learning-based CT fractional flow reserve assessment in acute chest pain: first experience. Cardiovasc Diagn Ther. 2020 Aug;10(4):820-830. doi: 10.21037/cdt-20-381. PMID 32968637
- [Background] Ma Q, Ma Y, Yu T, Sun Z, Hou Y. Radiomics of Non-Contrast-Enhanced T1 Mapping: Diagnostic and Predictive Performance for Myocardial Injury in Acute ST-Segment-Elevation Myocardial Infarction. Korean J Radiol. 2021 Apr;22(4):535-546. doi: 10.3348/kjr.2019.0969. Epub 2020 Nov 30. PMID 33289360
- [Background] Lee HC, Park JS, Choe JC, Ahn JH, Lee HW, Oh JH, Choi JH, Cha KS, Hong TJ, Jeong MH; Korea Acute Myocardial Infarction Registry (KAMIR) and Korea Working Group on Myocardial Infarction (KorMI) Investigators. Prediction of 1-Year Mortality from Acute Myocardial Infarction Using Machine Learning. Am J Cardiol. 2020 Oct 15;133:23-31. doi: 10.1016/j.amjcard.2020.07.048. Epub 2020 Jul 26. PMID 32811651
- [Background] Zheng Y, Li T. Letter to the Editor concerning the article "Machine learning for prediction of 30-day mortality after ST elevation myocardial infarction". Int J Cardiol. 2018 Sep 1;266:41. doi: 10.1016/j.ijcard.2017.11.061. No abstract available. PMID 29887469